CLINICAL TRIAL: NCT05101278
Title: Formation of Reactive Oxygen Species in Patients With Severe Traumatic Brain Injury in Normal vs Increased Oxygenation.
Brief Title: ROS in TBI Patients in Relation to Level of Oxygenation.
Acronym: ROS-TBI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: K2020-1148
Record Dates: First submitted 2021-10-06; First posted 2021-11-01 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Systemic Oxygenation vs ROS Formation in TBI Patients
Keywords: TBI, ROS, oxygenation, cerebral monitoring, neurointensive care
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and CSF samples for analysis of short-lived ROS and other markers of oxidative stress.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project an observational study performed on patients with severe Traumatic Brain Injury (TBI) treated at Neurosurgical ICU (NICU) at Karolinska University Hospital. The purpose of this study is to evaluate the effects of various oxygenation levels on production rate of Reactive Oxygen Species (ROS) in patients with severe traumatic brain injury (TBI). The patients will be included in the study after the placement of intracranial monitoring device consisting of intracranial pressure gage (Codman), microdialysis (MD), and Licox oxygen electrode for measurement of partial pressure of oxygen in brain tissue (pBtO2). Intracranial monitoring is inserted on clinical indications and is used for early detection of deleterious processes in brain tissue such as hypoxia or hypoperfusion and for purpose of guiding of given therapies such as cerebral perfusion pressure (CPP), oxygenation, dosage of vasoactive drugs etc. Despite the technical possibilities to monitor all these physiological parameters, there are no clear guidelines how to interpret the MD and pBtO2 data and implement it in clinical decision making. One of the controversies deals with optimization of oxygen levels: some authors point out the importance of adequate brain tissue oxygenation, whereas other researchers are worried about the possible negative effects of excessive oxygen levels such as increased production of ROS or facilitating pulmonary atelectasis, contributing to adverse outcome.

The purpose of this study is to investigate the effect of various oxygenation levels on ROS production in TBI patients.

This pilot study is designed to measure short-lived ROS in blood and microdialysis fluid samples of TBI patients during alternating periods of normal vs temporarily increased oxygenation levels under normobaric conditions (normal atmospheric pressure).

ELIGIBILITY:
Inclusion Criteria:

1. Severe isolated TBI (GCS<8, AIS =<3), CT-verified TBI (tSDH,tEDH, tSAH, contusion bleedings) caused by blunt or penetrating trauma.
2. Established intracranial monitoring (ICP, MD, LiCox pBtO2) at NICU.
3. Age >= 18
4. Time from trauma from 0 to 4 days.
5. Informed consent from Close relative.
6. Systemic hyperoxygenation can be used in patients with pBtO2 <20 mmHg, based on clinical decision.

Exclusion Criteria:

1. Major extracranial injury, AIS >3
2. Brain dead or expected survival <24 hours
3. Pregnancy
4. Respiratory insufficiency FiO2> 40%

6. No consent from relative.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe isolated TBI with established intracranial monitoring (based on clinical desision), inclusion between 0 to four Days from their injury.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ROS concentrations in blood | 7 days
  ROS concentrations in patient´s blood will be measured repeatedly at normal systemic oxygenation and at increased oxygenation if necessary.
Markers of oxidative stress | 7 days
  Indirect markers of oxydative stress, as MDA (Malondialdehyde) and Isoprostane F2, in relation to level of systemic oxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden